CLINICAL TRIAL: NCT04461587
Title: Examination of Pirfenidone (Esbriet®) Therapy in Coal Workers' Pneumoconiosis With Pulmonary Fibrosis Associated With Radiographic and Functional Impairment to Examine the Reduction in Progression of Disease, Reduction of Exacerbation Rates and Possible Reduction of Inflammatory Biomarkers as an Index of Clinical Response.
Brief Title: Examination of Pirfenidone (Esbriet®) Therapy in Coal Workers' Pneumoconiosis With Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmonary Research of Abingdon, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42227
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Coal Workers' Pneumoconiosis (Complicated)
Keywords: Black Lung; Black Lung Disease; Coal Miner's Lung; Coal Worker's Pneumoconiosis; Coalworker's Pneumoconiosis; Pneumoconiosis, Coal Worker's
MeSH Terms: conditions — Anthracosis | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: Open label interventional study observing US FDA approved Esbriet (for Interstitial Pulmonary Fibrosis) in Coal Workers' Pneumoconiosis patients with pulmonary fibrosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pirfenidone [Esbriet] (Experimental): Pirfenidone recommended daily dose for patients is 801 mg three times a day with food, for a total of 2403 mg/day. Upon initiating treatment, the dose should be titrated to the recommended daily dose of 2403 mg/day over a 14day period as follows:
  * Days 1 to 7: a dose of 267 mg administered three times a day (801 mg/day)
  * Days 8 to 14: a dose of 534 mg administered three times a day (1602 mg/day)
  * Day 15 onward: a dose of 801 mg administered three times a day (2403 mg/day) It will be provided in 267mg capsules. Treatment will be for a minimum of 12 months. Treatment duration will continue until last patient enrolled received 12 months of treatment.
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — see previous entries
  Other Names: Esbriet

SUMMARY:
Examination of pirfenidone (Esbriet®) therapy in coal workers' pneumoconiosis (black lung) with pulmonary fibrosis (scarring of the lung).

DETAILED DESCRIPTION:
Examination of pirfenidone (Esbriet®) therapy in coal workers' pneumoconiosis with pulmonary fibrosis associated with radiographic and functional impairment to examine the reduction in progression of disease, reduction of exacerbation rates and possible reduction of inflammatory biomarkers as an index of clinical response.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to provide informed consent and to comply with study protocol
* 2. Coal miners between the ages 40 to 79 years of age at visit 1with a minimum of 15 years in a coal mining environment
* 3. Chest CT Scan or Chest Xray (within 6 months) confirming diagnosis of CWP, complicated black lung disease/progressive massive fibrosis will be recorded. If CT not available must be obtained at Visit 1.
* 4. Evidence of Loss of lung function defined by decline in FEV1 or FVC or DLCO of 5% within the past 36 months prior to enrollment.
* 5. FEV1 ≤ 75% or FVC ≤ 80% or DLCO ≤ 70% or abnormal 6MWT with oxygen desaturation of 4% or greater than resting at screening or within past 6 months.
* 6. Former smokers and current smokers will be enrolled if documented evidence of CWP/PMF is present and meet PFT guidelines. Current smokers will be given smoking cessation counseling at each visit due to the effect on pirfenidone concentration and efficacy.

Exclusion Criteria:

* 1. History of prior therapy with Esbriet or Ofev (pirfenidone or nintedanib)
* 2. Recent hospitalization (within 30 days prior to screening) for respiratory decompensation.
* 3. Patients using monoclonal antibody therapy or immunosuppressive therapy for other disease process will be excluded, except for the following:

  * Daily prednisone up to 10 mg daily (prescribed for lung disease or rheumatoid arthritis) will be permitted. Chronic use for 3 months prior to enrollment will be documented.
  * Methotrexate for rheumatoid arthritis will be permitted as long as chronic use for 6 months prior to enrollment is documented.
* 4. Elevation of liver function test at screening documenting AST, ALT or total bilirubin > 3 x ULN or ALP > 2.5 x ULN.
* 5. Patients who have other pulmonary pathology such as lung cancer, active tuberculosis or atypical mycobacterial infection requiring treatment.
* 6. Patients with recurrent malignancy requiring chemotherapy or radiation therapy. Individuals with a prior diagnosis of localized skin cancer, prostate cancer, localized bladder cancer will not be excluded unless undergoing active treatment. Patients with a prior diagnosis of malignancy treated greater than 5 years ago will be considered for enrollment.
* 7. History of alcohol or drug abuse that would impair or risk the patient's full participation in the drug study in the opinion of the investigator
* 8. Use of any investigational therapy within 4 weeks of enrollment.
* 9. Individuals with clinically significant unstable cardiac disease (ejection fraction ≤35%) or complex arrhythmias per PI discretion. Chronic atrial fibrillation will be permitted if heart rate is controlled. Historical values of ejection fraction will be accepted.
* 10. Individuals with poorly controlled diabetes per PI discretion (Hemoglobin A1c >9). Historical values will be accepted.
* 11. Pregnancy or lactation.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 12 months minimum
  Primary objective for this study is to determine the rate of decline ( relative change in FVC (% and ml) in patients with coal workers' pneumoconiosis (Black Lung) with pulmonary fibrosis (CWP/PMF) during treatment with pirfenidone (Esbriet®).

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 12 months minimum
  rate of decline (relative change in % and ml )of FEV1 compared to baseline assessments established at enrollment.
Diffusing capacity of the lung for carbon monoxide (DLCO) | 12 months minimum
  rate of decline (relative change in %) of DLCO compared to baseline assessments established at enrollment.
6 minute walk test | 12 months minimum
  rate of decline of 6 minute walk test compared to baseline assessments established at enrollment.
Chest CT | 12 months
  Chest CT scans will be reviewed to determine if radiographic progression occurs during therapy.
Inflammatory biomarkers | 12 months minimum
  The reduction of inflammatory biomarkers (Interleukin-6 [IL-6], Transforming Growth Factor Beta 1 [TGF-β 1] and Tumor Necrosis Factor Alpha [TNF-α]) and the potential reduction correlation with change in lung function
St. George's Respiratory Questionnaire (SGRQ) | 12 months minimum
  Change in total score compared to baseline. Total score summarizes the impact of the disease on overall health status. Scores range from 0 - 100, with higher scores indicating more limitations.

OTHER OUTCOMES:
Rates of Respiratory Exacerbation | 12 months minimum
  Change in exacerbation rate compared to 12 months prior to enrollment, including respiratory-related hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Emory Robinette, MD, Principal Investigator — Pulmonary Research of Abingdon, LLC
Locations (1):
- Pulmonary Research of Abingdon, LLC, Abingdon, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: European Journal of Respiratory Medicine Journal Article — https://europeanjournalofrespiratorymedicine.com/pirfenidone-therapy-in-coal-workers-pneumoconiosis-with-pulmonary-fibrosis-and-associated-functional-impairment